CLINICAL TRIAL: NCT03579238
Title: Entrainment Interaction Between Physician and Patient During Palpation of the Cranium
Brief Title: Entrainment Between Clinician and Patient During Palpation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Michael Seffinger, Professor, Western University of Health Sciences
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1209771-1
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Doctor Patient Relation
MeSH Terms: interventions — Touch

STUDY DESIGN:
Intervention Model Description: Intrasubject sequential intervention design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinicians, participants, researchers and statistician will not know which stage of interaction (distant, close, touching, pulling) induces entrainment, if at all. Statistician will be blinded to stage allocation of each data set, and stages of interaction will be randomized per encounter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Distant (No Intervention): The clinician sits quietly 3 feet away from participant who is lying on a soft table at rest.This position is held for 5 minutes without moving.
- close (No Intervention): The clinician sits at the head of the table with his arms on the table alongside the participant's head but not touching the resting patient who is lying at rest on the table. This position is held for 5 minutes without moving.
- touching (Sham Comparator): The clinician lifts the patient's head passively off the table in order to place his hands underneath the participant's head, palms facing upwards and in contact with the back of the head of the participant. The participant's head is gently lowered to rest upon the clinician's hands. No external force is provided by the clinician upon the participant's head as the head rests in the clinician's palms on the table. This position is held for 5 minutes without moving. This is called a "touching" intervention and is meant to be a sham. A five minute rest period follows in which the clinician removes his hands from underneath the participant's head and places them next to the patient on the table, but not in contact with the patient.
  Interventions: Procedure: touching
- Occipital motion inhibition (Experimental): The clinician gently inhibits motion of the participant's occiput into flexion phase of the primary respiratory mechanism, and allows extension phase only. Upon sensing a still point, where no further flexion motion is palpated, the clinician will state to the research assistant "now" to indicate he feels a still point. This position is held for 5 minutes without moving. This is called a CV4 or modified CV4 intervention. A five minute rest period follows in which the clinician removes his hands from underneath the participant's head and places them next to the patient on the table, but not in contact with the patient.
  Interventions: Procedure: CV4

INTERVENTIONS:
Procedure: CV4 — The occiput of a supine patient is held such that flexion motion is inhibited and extension motion is reinforced.
  Other Names: Modified CV4, CV-4
  Arms: Occipital motion inhibition
Procedure: touching — the clinician allows the participant's head to rest quietly upon his open palms on a table.
  Other Names: light touch
  Arms: touching

SUMMARY:
This study will assess the physiological interaction between the palpating clinician and a research participant using a laser Doppler flow meter to detect changes in blood flow parameters.

DETAILED DESCRIPTION:
Research participants will lie on their backs on a soft table while a licensed physician, with special training in osteopathic palpation and manipulation approaches, touches, and administers a slight inhibition of occipital bone motion for five minutes per stage. Both will have a non invasive skin sensor (probe), called a laser Doppler flow meter, attached to their forehead to detect changes in subcutaneous blood flow velocity. The signal from the device will be augmented and transmitted for display onto a digital polygraph recorder. Then, using Fourier transformation software, the signal will be displayed as a graph for spectral analysis to determine the effect on specific wave forms related to autonomic activity. The interaction between the two individuals will be assessed for evidence of entrainment phenomenon, i.e., the influence of one biorhythm upon another.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult that can lie on his or her back on a padded table without moving for 35 minutes.

Exclusion Criteria:

* head trauma within the last six months, seizure disorder, pregnant, brain disease or injury, using beta or alpha blocker medication, unable to lie still for 35 minutes, allergy to the hypoallergenic sticky tape used to attach sensor to forehead

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Entrainment of still points between clinician and research participant | within 1 minute of each other (arbitrary designation)
  When one person has a still point it may or may not affect the other person. If it does, then entrainment will have occurred. The clinician's intent is to create a still point in the participant by inhibiting occipital motion. This is measurable using the laser Doppler flow meter. The induction of the still point, which is manifest on the polygraph and in spectroscopy as a distinct diminished amplitude at the .08-1.5 Hz frequency, may entrain the clinician to have a still point as well.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seffinger, D.O., Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No
The overall results of the study and examples of entrainment phenomenon can be extracted from the data gathered for sharing and informational purposes.